CLINICAL TRIAL: NCT01487135
Title: A Randomized, Double-blind, Placebo- and Active-controlled, 3-way Crossover, Phase 1 Study to Evaluate the Effect of EVP-6124 at Therapeutic and Supratherapeutic Concentrations Following a 2-dose EVP-6124 Regimen on the QT Interval in Healthy Male and Female Subjects.
Brief Title: Phase 1 Study to Assess the Effects of EVP-6124 on the QT/QTc Interval in Healthy Subjects
Acronym: TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EVP-6124-012
Record Dates: First submitted 2011-11-29; First posted 2011-12-07 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Subjects; Cardiac Repolarization
Keywords: Thorough QT (TQT); EVP-6124
MeSH Terms: interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EVP-6124 (Experimental): A single low dose of 8-mg EVP-6124 and A single high dose of 80-mg EVP-6124
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): Cranberry juice (180 mL)
  Interventions: Drug: EVP-6124
- Moxifloxacin (Active Comparator): A single dose of 400-mg Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: EVP-6124 — A single oral low dose of EVP-6124 in cranberry juice (180 mL) administered on Day 1 and a high dose of EVP-6124 in cranberry juice (180 mL) administered on Day 2.
  Arms: Placebo
Drug: Placebo — Cranberry juice only (180 mL) administered orally on both Day 1 and Day 2.
  Arms: EVP-6124
Drug: Moxifloxacin — A moxifloxacin 400 mg tablet administered orally on Day 1
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the effect of EVP-6124 at therapeutic and supratherapeutic concentrations on cardiac repolarization in healthy subjects.

DETAILED DESCRIPTION:
Subjects will be randomized to six treatment sequences of 10 subjects each. Subjects will be admitted to the clinic on Day -1 before dosing. Each of the EVP-6124 and placebo treatment periods (blinded) will include a 10-day/9-night confinement to the Clinical Pharmacology Unit (CPU) with study drugs being administered on Day 1 and Day 2. The moxifloxacin treatment period (open-label) will include a 3-day/2-night confinement to the CPU with moxifloxacin administration on Day 1.

The study will include 2 washout periods in which each washout starts from the time of the last dose of the preceding treatment period to the first dose of the next treatment period. The washouts following the EVP-6124 or placebo treatments will be 30 days while the washout following the moxifloxacin treatment will be 7 days. Follow-up visit (5 to 10 days following discharge from the CPU).

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc for 60 days prior to the administration of the study medication)
* Physically and mentally healthy volunteers

Exclusion Criteria:

* Clinically significant electrocardiographic abnormality in the opinion of the Investigator
* History of cardiovascular abnormalities/conditions including syncope in the 3 months preceding enrollment or any history of significant previous cardiac arrhythmia;
* Potassium levels outside of the normal ranges (3.5 to 5.2 mEq/L)
* Clinically significant deviations from normal blood pressure (BP) as judged by the Investigator
* Currently have, or have a history of, disease or dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system, that is clinically significant in the opinion of the Investigator
* Unwilling to refrain from strenuous exercise from 3 days prior to baseline Day -1 through discharge of each treatment period
* Family history of Torsade de Pointes or long-QT syndrome, or cardiac death or sudden death without a preceding diagnosis of a condition that could be causative of sudden death
* Evidence of any chronic medical condition requiring prescription medications
* History of study drug allergy (including moxifloxacin, likely hypersensitivity or allergies to EVP-6124, or any components of EVP-6124)
* Current or history of drug or alcohol abuse within the past year
* Abnormal preadmission clinical laboratory evaluations which are considered clinically significant by the Principal Investigator
* Any subject considering or scheduled to undergo any surgical procedure during the study
* Acute illness within 7 days prior to study agent administration or have had a major illness or hospitalization within 1 month prior to study agent administration
* Any subject who has received any known hepatic or renal clearance altering agents within 30 days prior to the first dose of study drug
* A positive serology test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody at screening
* A positive urine drug screen for ethanol or substances of abuse including cocaine,cannabinoids, phencyclidine, amphetamines, benzodiazepines, barbiturates, opiates, propoxyphene, and methadone at check-in(s)
* Female subjects of childbearing potential with positive serum pregnancy test at screening or baseline (Day -1) of each treatment period. Sexually active females who refuse to take appropriate steps not to become pregnant during the course of the clinical study
* Men, sexually active with female partners of childbearing potential, who are unwilling to use appropriate contraception during the course of the study and for 30 days after discharge from the last treatment period
* Donated plasma or blood within 30 days prior to the first dose of study medication or has a history of blood donation of more than 450 mL within 3 months prior to dosing
* Use of any prescription medications/products, within 14 days prior to dose administration on Day 1 of Treatment Period 1, unless deemed acceptable by the Investigator
* Use of any over-the-counter, nonprescription preparations (including minerals, and phytotherapeutic/herbal/plant-derived preparations), within 14 days prior to dose administration on Day 1 of Treatment Period 1, with the exception of acetaminophen used at recommended doses
* Use of investigational drug 30 days prior to Day -1 of Treatment Period 1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change-from-baseline in individual corrected QTc (ΔQTcI) for EVP-6124 vs. placebo | Day 1: predose to 20 hours postdose; Day 2 predose to 168 hours postdose
  Change-from-baseline in Fridericia's correction QTc (ΔQTcF) and change-from-baseline in Bazett's correction QTc (ΔQTcB) will be secondary variables.
  The placebo-corrected baseline-adjusted QTc (ΔΔQTc), calculated as differences between time-matched mean change-from-baseline QTc values obtained on Day 1 (low dose) and on Day 2 (high dose) of the EVP-6124 treatment relative to the corresponding QTc values obtained on Day 1 and Day 2 of the placebo treatment, will be evaluated to quantify the effect of EVP-6124 on cardiac repolarization.

SECONDARY OUTCOMES:
Change-from-baseline in individual corrected QTc (ΔQTcI) for positive control vs. placebo | Day 1: predose to 20 hours postdose
  The placebo-corrected baseline-adjusted QTc (ΔΔQTc), calculated as differences between time-matched mean change-from-baseline QTc values obtained on Day 1 of the moxifloxacin treatment relative to QTc values obtained on Day 1 of the placebo treatment, will be evaluated to establish assay sensitivity.
Safety and tolerability of EVP-6124 at low dose and high doses | Day -1 through follow-up (5 to 10 days after discharge)
  All AEs (adverse experiences) spontaneously reported by subjects and/or observed by investigator and evaluation of physical examinations, prior and concomitant medications, clinical laboratory tests, ECGs, and vital signs measurements.